CLINICAL TRIAL: NCT05683795
Title: Pathophysiology, Mitigation, and a Core Outcome Set for the Empty Pelvis Syndrome After Pelvic Exenteration: a Delphi-study by the PelvEx Collaborative
Brief Title: PelvEx - Beating the Empty Pelvis Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: ERGO: 77306
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Empty Pelvis Syndrome; Pelvic Exenteration; Pelvic Neoplasm; Pelvic Cancer; Rectal Cancer; Postoperative Complications
Keywords: Empty Pelvis Syndrome; Pelvic Exenteration
MeSH Terms: conditions — Pelvic Neoplasms; Rectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Professionals: Members of The PelvEx Collaborative who are experts in performing pelvic exenteration surgery, and managing the complications relating to the empty pelvis syndrome as a result of this surgery.
  Interventions: Other: Consensus study
- Patient Representatives: Patients that have undergone pelvic exenteration surgery and likely to have been exposed to the morbidity of the empty pelvis syndrome.
  Interventions: Other: Consensus study

INTERVENTIONS:
Other: Consensus study — Modified-Delphi study and consensus meetings

SUMMARY:
The empty pelvis syndrome is an unsolved and poorly defined problem severely affecting patients that have pelvic exenteration surgery, and also the teams looking after them. It is unclear what the anatomical and pathophysiological causes of the empty pelvis syndrome are, how it can be prevented, and how its sequelae can be measured. The evidence to guide decisions around the empty pelvis syndrome is of low quality, and so there is a large amount of variation in approaches between different hospitals.

This consensus study will define a core outcome set for the empty pelvis syndrome, and establish current levels of consensus on pathophysiology and mitigation of the empty pelvis syndrome through a modified-Delphi process involving both healthcare professionals and patient representatives.

DETAILED DESCRIPTION:
Rationale for a consensus study:

A measurable core outcome set for the empty pelvis syndrome will allow more directed research in this area. A core outcome set specifies a minimum set of outcomes to be measured for a particular health issue. Core outcome measures standardise and reduce bias in research. Selection of appropriate outcomes is essential in designing trials so that different treatments can be compared directly and efficiency, and therefore research in a particular area is improved. The Core Outcome Measures in Effectiveness Trials (COMET) database was searched on 14/07/2022 and there were no references to pelvic exenteration, complex pelvic cancers or the empty pelvis syndrome. Outcomes need to be relevant and important to stakeholders in a given problem, in the case of the empty pelvis syndrome this includes both patients and healthcare professionals. The study protocol presented here endeavours to address this gap in the literature, and has had involvement of patient representatives in its design.

In order to define and develop a core outcome set for the empty pelvis syndrome a modified-Delphi study is proposed. In addition to this consensus on the pathophysiology of the empty pelvis syndrome and which preventative reconstructive surgical techniques will be investigated.

The Expert Groups:

This Delphi study has been designed through The PelvEx Collaborative in accordance with the Guidance on Conducting and Reporting Delphi Studies (CREDES) guidelines, and The COMET Handbook. In order to undertake a Delphi study a panel of experts are required. The PelvEx Collaborative is a diverse international group of health care professionals from 140 hospitals across five continents that provide pelvic exenteration services, and aim to improve the results for patients after pelvic exenteration surgery. This is an ideal, motivated and logistically convenient platform to undertake a Delphi study due to its rich healthcare professional expert group and its access to patients as key stakeholders. In a Delphi study there is no agreement on how a group of experts should be selected, and there is no need for a statistically representative sample to be obtained. Therefore, all members of The PelvEx Collaborative will be invited to be involved in the study, generating, multi-professional, multi-national representation.

The PelvEx Collaborative are experts in providing complex pelvic cancer treatment, however they are not experts in actually undergoing pelvic exenteration and suffering the complications of the empty pelvis syndrome. Patients are essential stakeholders, so in accordance with COMET patient involvement from an early stage has been sought in the design of this project. Patient representatives will be recruited through colleagues in The PelvEx Collaborative, Bowel Research UK Patients and Researchers Together (BRUK PaRT), CommunitiesFirst, and the World Federation of Incontinence and Pelvic Problems (WFIPP). For non-English speaking patients representatives that would like to take part, participating members of The PelvEx Collaborative will be required to assist in the translation of statements from English, professional translation services may also be sought to facilitate this process.

The Delphi Pilot Process (Completed December 2023):

A modified-Delphi study will be performed. The systematic review (Johnson et al.) and subsequently published literature on the empty pelvis syndrome was used to formulate pilot statements for voting, which were supplemented with formal and informal discussions from PelvEx 2022. A project steering committee was formed to include multi-national representatives from The PelvEx Collaborative, and patient representatives. Discussions with the steering committee further informed Delphi statements, the steering committee then completed a pilot of the first round of the Delphi.

Pilot statements were divided into three domains - an empty pelvis core outcome set, pathophysiology of the empty pelvis syndrome, and mitigation of the empty pelvis syndrome. These were scored from 1 - 9 on a Likert scale, as recommended by the Grading of Recommendations Assessment, Development and Evaluation (GRADE) working group. With 1-3 representing 'not important', 4-5 representing 'important but not critical' and 7-9 representing 'critical for inclusion.' It was also decided to include '0' on the scoring, which represented 'unable to comment.'

Following discussions within the steering committee it was decided that patient representatives would not take part in voting on pathophysiology or mitigation of the empty pelvis, as they would be unlikely to have the experience in this area to provide helpful input into forming a consensus. All statements in each domain were arranged in alphabetical order to reduce leading questions or researcher bias. The final question on each domain was an open question in order to avoid early closure of ideas among participants so that further insight that had not been anticipated from the literature could be gained.

Following completion of the piloting process the results were reviewed by the steering committee, who then met to discuss presentation of results, revisions, additional final statements, a priori consensus and dissemination of the Delphi study. Once this pilot testing was completed, the protocol will be published onto the COMET database to ensure transparency of reporting.

First Delphi Round (Anticipated start in January 2023):

Participants will be given one month to complete questionnaires with email reminders at 2 weeks, and 48 hours from the deadline. To encourage responses reminder emails will be personalised and will give information on questionnaire completion rates. Any participants that wish to drop out will be encouraged to give a reason for doing so in order to make recognition of any attrition bias easier to detect.

In order to be able to describe the diversity of expert groups demographic information will also be requested, this will not include special category data defined under General Data Protection Regulation and the Data Protection Act 2018.

The completed pilot-Delphi will be disseminated and data collected using the Qualtrics survey software. The first round of the Delphi will include the piloted open questions for the reasons given above, subsequent Delphi rounds will not include open questions.

First-round analysis:

Analysis and presentation of patient representative and healthcare professional data will take place separately. It is anticipated that there will be far more healthcare professionals in the study, therefore attempting to analyse these two groups together will reduce the importance given to the patient voice.

There is no recognised formal way of defining consensus in Delphi studies, however it is specified here a priori that in order for statements to progress they must obtain stricter consensus between subsequent rounds, based on the work of Blazeby et al. To progress from the first round to the second round statements must be rated 7 - 9 by 50% or more of participants, and by 1 - 3 by no more than 15% of participants in at least one stakeholder group. Beyond round 2 retained items must be rated between 7 - 9 by over 70% of respondents, and by 1 - 3 by less than 15% by at least one stakeholder group. This method reduces the chance of dropping statements that may have been rated more highly in subsequent rounds once participants have received feedback. From piloting there was concern that a large proportion of statements for the core outcome set were rated as essential, therefore the steering committee decided a priori that if there are 10 or more core outcome set statements reaching consensus by the end of a second round then a third Delphi round will take place with higher levels consensus required, defined as 95% participants voting 7 - 9 that the statement should be included, this is line with Innes et al.

Responses to open questions will undergo thematic analysis and will be used to formulate new statements for addition to subsequent rounds. Any comments that apply to particular statements, that are not able to be formulated into new statements will be presented verbatim in subsequent rounds alongside relevant statements. Further qualitative information will not be sought after round 1.

Responses will be analysed and presented separately for healthcare professionals and patient representatives using medians and interquartile ranges. This is preferred to means and standard deviations to reduce the effect of outlier responses. Histograms will also be included to help patient representatives that are unfamiliar with descriptive statistics understand the results.

Subsequent rounds:

Only individuals that completed the previous round will be contacted to take part in a subsequent round. The same timelines will apply for subsequent rounds, with invitations to take part presented as a personal email to the participant with a report on response rates from around the world to encourage ongoing involvement. New statements generated from thematic analysis will be added, again placed in alphabetical order with the others. It will be reiterated to participants that the aim is to achieve consensus, and participants will be invited to re-consider their previous responses but will be under no obligation to do so.

Subsequent analysis:

It is anticipated that there will be 3 rounds of questionnaires, it is possible there may be a requirement for more rounds, however this will depend on attrition, consensus and stability of consensus. The Delphi may stop earlier if a strict consensus has been reached on all statements. These decisions will be made by the Delphi study committee once analysis has taken place. Analysis will take place in the same manner between each round with median, interquartile range, histogram and a check of consensus.

If attrition drops to below 70% of a previous round the Delphi study will be terminated, as below this level rigour cannot be guaranteed. Attrition analysis will be undertaken between rounds to assess whether systematic attrition bias is occurring. Participants dropping out of the study will be encouraged to give reasons for dropping out in order to supplement this analysis.

Consensus meetings:

Following completion of the final Delphi round final consensus meetings will take place. For statements from the first domain (core outcome set) for the empty pelvis syndrome, any statements that have reached consensus or possibly may reach consensus at face-to-face meetings will have options of instruments measuring for outcomes prepared in accordance with COnsensus-based Standards for the selection of health Measurement Instruments (COSMIN)/COMET guidance. This will allow definition of both what to measure for the empty pelvis syndrome and how to measure it, therefore reducing the need for subsequent consensus meetings.

It is anticipated that the majority of the core outcome set will be straightforward to measure. For aspects of the core outcome set that are more difficult to measure all potential instruments for measurement will be selected using the expert opinion of the project steering committee and reviews of the relevant literature. This will include instrument feasibility assessments. These options will then be presented at consensus meetings.

PelvEx 2023 is the international meeting of The PelvEx Collaborative and is an ideal time to hold a face-to-face consensus meeting for participating healthcare professionals, the meeting is currently due to go ahead in France in July 2023. It is an opportunity to capture a global audience in an environment where audience participation and voting already happens as a matter of course. It was felt that this meeting, however, would not be appropriate for patient representatives as it will involve significant travel, and will need to be fitted into an academic timetable. Moreover, patients may be heavily influenced by the opinions of healthcare professionals, and they may not feel as able to voice their opinions in front of a large audience.

To increase the number of involved patient representatives, give them the time they need to consider statements, and provide a less intimidating environment it is planned to hold virtual consensus meetings prior to PelvEx 2023. Beforehand patients will be sent results from the final round of Delphi, including how they have voted. If non-English speaking patient representatives wish to take part then appropriate multi-lingual healthcare professionals will need to be present to assist with translation. Participants will be asked to complete some demographic information to allow diversity reporting. Any statements retained from previous Delphi rounds for the core outcome set will be included and participants will be asked to vote on whether they should stay in, be removed, or whether they are unsure. Where there is no consensus or participants are unsure then further discussion will take place, also considering whether statements overlap and can be combined. Further voting will take place, followed by further discussion, if there is persistent disagreement a final round of voting will take place using a majority rule.

For the core outcome set statements felt to be important to be included possible instruments to measure these statements will be presented for approval. It is anticipated that selection of instruments for patients will be difficult as the evidence on their methodology is likely to be difficult to understand, however it is hoped that with support from research facilitators that patients will be able to judge relevance, comprehensiveness and comprehensibility of the available outcome instruments. This meeting will be recorded for analysis and potential presentation of patients speaking at PelvEx 2023 to help healthcare professionals understand the patient experience.

Prior to PelvEx 2023 the results of the final Delphi rounds, statements for voting, and the patient virtual consensus meeting will be sent out to participating healthcare professionals, including how individuals that participated previously voted. A list of delegates will be obtained along with their institutions to allow reporting of the diversity of the audience, this will also include whether or not participants were involved with the Delphi study itself. The presentation given will include a brief overview of this information, before progressing onto voting on any statements that have progressed from the final Delphi round. As per the patient representative consensus meeting voting will take place as either yes, no, or unsure. If consensus is not reached on a particular topic then further discussion will take place where an effort will be made to capture dissenting views to determine the nature of a polarised response. A further round of voting will take place, if no consensus is reached then there will be further discussion, and finally voting by a majority rule. Statements that are felt to be overlapping may be combined. Again, for the core outcome set domain, statements that have reached consensus will also have their valid options for their instruments to measure them presented in accordance with COSMIN/COMET guidance. This will reduce the need for future consensus meetings. If there is only one possible instrument to use then this will be presented with a decision on yes or no.

It is difficult to predict how many statements will require voting and discussion at the meeting, and whether there will be time to discuss instruments for measuring a core outcome set. A further round of voting, or a virtual meeting following PelvEx 2023 after face-to-face discussions may be required and this will be at the discretion of the project steering committee.

Reporting of results:

Reporting of results will be using Core Outcome Set-STAandards for Reporting (COS-STAR) Guidelines. Any deviations from the above protocol will be described and justified. In addition statements from the third domain, which describe treatment options to reduce the effects of the empty pelvis syndrome, will be graded by strength of recommendation and level of evidence according to two predefined scales proposed by the European Association for Cardio-Thoracic Surgery clinical guidelines.

Once the process described above has been completed a final draft of the results of the project will be reviewed by an external board prior to publication and dissemination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare professional and member of The PelvEx Collaborative
2. Patient representative that has undergone pelvic exenteration surgery - defined as surgery to remove multiple organs from the pelvis, including beyond total mesorectal excision plane operations, for any pelvic malignancy (i.e., primary or recurrent colorectal, gynaecological, urological, and connective tissue disease)
3. Non-English speaking healthcare professionals and patient representatives where language translation is possible.

Exclusion Criteria:

1. Patient representatives that have not undergone pelvic exenteration surgery.
2. Non-English speaking healthcare professionals and patient representatives where language translation is not possible.
3. Individuals unable to take part in the online consensus process, or unable to give online consent digitally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An international cohort of patients that have undergone pelvic exenteration surgery, and an international group of expert clinicians who perform pelvic exenteration surgery (The PelvEx Collaborative).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
A core outcome set for the empty pelvis syndrome | 8 months
  Consensus process involving both healthcare professionals and patient representatives to define measurable outcomes for the empty pelvis syndrome

SECONDARY OUTCOMES:
Consensus on pathophysiology of the empty pelvis syndrome | 8 months
  Process to establish where there is consensus on the pathophysiology for the empty pelvis syndrome among healthcare professionals
Consensus on mitigation of the empty pelvis syndrome using reconstructive techniques | 8 months
  Process to establish where there is consensus on the reconstructive techniques to mitigate the effects of the the empty pelvis syndrome among healthcare professionals

CONTACTS AND LOCATIONS:
Overall Officials: Charles T West, MBBS BSc, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of University of Southampton, between Delphi rounds identifiable information will be anonymised and non-attributable to participants. Anonymised or statistical data may be used publicly or shared with third parties.

REFERENCES:
- [Background] Johnson YL, West MA, Gould LE, Drami I, Behrenbruch C, Burns EM, Mirnezami AH, Jenkins JT. Empty pelvis syndrome: a systematic review of reconstruction techniques and their associated complications. Colorectal Dis. 2022 Jan;24(1):16-26. doi: 10.1111/codi.15956. Epub 2021 Oct 25. PMID 34653292
- [Background] Sutton PA, Brown KGM, Ebrahimi N, Solomon MJ, Austin KKS, Lee PJ. Long-term surgical complications following pelvic exenteration: Operative management of the empty pelvis syndrome. Colorectal Dis. 2022 Dec;24(12):1491-1497. doi: 10.1111/codi.16238. Epub 2022 Jul 19. PMID 35766998
- [Background] Blazeby JM, Macefield R, Blencowe NS, Jacobs M, McNair AG, Sprangers M, Brookes ST; Research Group of the Core Outcomes and iNformation SEts iN SUrgical Studies-Oesophageal Cancer; Consensus Group of the Core Outcomes and iNformation SEts iN SUrgical Studies-Oesophageal Cancer. Core information set for oesophageal cancer surgery. Br J Surg. 2015 Jul;102(8):936-43. doi: 10.1002/bjs.9840. Epub 2015 May 18. PMID 25980524
- [Background] Innes K, Hudson J, Banister K, Croal B, Ramsay C, Ahmed I, Blazeby J, Gillies K; CGALL Trial Group. Core outcome set for symptomatic uncomplicated gallstone disease. Br J Surg. 2022 Apr 5:znac095. doi: 10.1093/bjs/znac095. Online ahead of print. PMID 35381067
- [Derived] PelvEx Collaborative. Beating the empty pelvis syndrome: the PelvEx Collaborative core outcome set study protocol. BMJ Open. 2024 Feb 5;14(2):e076538. doi: 10.1136/bmjopen-2023-076538. PMID 38316595